CLINICAL TRIAL: NCT03816566
Title: Validation of a Wearable Non-invasive Device (the Patch) to Aid in Diagnosing Sleep Apnea
Brief Title: Validation of a Wearable Non-invasive Device (the Patch)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: BresoTEC Inc. (Industry)
Responsible Party: Sponsor
Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: CL-00001
Record Dates: First submitted 2019-01-23; First posted 2019-01-25 (Actual); Last update posted 2019-01-25 (Actual); Status verified 2019-01

CONDITIONS: Sleep Apnea
MeSH Terms: conditions — Sleep Apnea Syndromes | interventions — Transdermal Patch

STUDY DESIGN:
Masking Description: The outcome assessor performing the automatic analysis of the patch data will be blinded to the PSG scores performed by the Sleep Lab Technicians.
  The principal investigator responsible for the completion and closing of the study according to the protocol will be blinded to the patch AHI automatic analysis.
  Similarly, the Sleep Lab Technicians scoring the PSG will be blinded to the patch automatic analysis.
  By the end of recruiting the target sample size, the data will be un-blinded and statistical analysis will be performed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Wearable Device and PSG (Experimental): The device under investigation (the patch) will be used in patients undergoing overnight polysomnography simultaneously, to compare the accuracy of the investigational device against the gold standard for the diagnosis of sleep apnea.
  Interventions: Device: patch

INTERVENTIONS:
Device: patch — A standalone wearable device (the patch), that can record tracheal sounds with a microphone attached just above the suprasternal notch of the subject. The patch also has a 3-dimensional accelerometer to record body position. Furthermore, the patch records oxygen saturation using an FDA cleared pulse oximeter, Nonin 3150 WristOx2® with Bluetooth Low Energy.

SUMMARY:
BresoTEC has designed and developed a standalone wearable device (the patch), that can record tracheal sounds with a microphone attached just above the suprasternal notch of the subject.

DETAILED DESCRIPTION:
The patch also has a 3-dimensional accelerometer to record body position. Furthermore, the patch records oxygen saturation using an FDA cleared pulse oximeter, Nonin 3150 WristOx2® with Bluetooth Low Energy. We have developed advanced signal processing algorithms to detect apneas and hypopneas. Many of these techniques for analyzing breathing sounds and detecting apneas and hypopneas have been published in peer-reviewed journals.

The goal of this study is to validate the patch against polysomnography (PSG) for use as an aid in the diagnosis of sleep apnea for adult patients. Our primary objective is to assess whether the estimated apnea-hypopnea index (AHI) calculated by the patch agrees with the results of an in-laboratory PSG.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria are men and women 18 years and above, who are referred to either the University Health Network (UHN), Toronto Rehabilitation Institute (TRI) or Toronto General Hospital sleep laboratories for overnight PSG because of a suspicion of a sleep disorder. It is intended for the general outpatient population.

Exclusion Criteria:

* Exclusion criteria are patients with suspected complicated co-morbidities including in-hospital patients and those who self-report diagnosis of heart failure, recent stroke, neuromuscular disorders, renal failure, obesity hypoventilation, COPD, or other severe lung diseases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-12-23 (Actual); Primary Completion 2019-08-23 (Estimated); Study Completion 2019-08-23 (Estimated)

PRIMARY OUTCOMES:
Estimation of AHI | 8 months
  Validate the performance of the patch in estimating the AHI compared to an in-laboratory PSG.

SECONDARY OUTCOMES:
Estimation of body position | 8 months
  Validate the performance of the patch in estimating body position during sleep compared to an in-laboratory PSG.

CONTACTS AND LOCATIONS:
Overall Officials: Clodagh Ryan, MD, Principal Investigator — Toronto General Hospital & Toronto Rehabilitation Institute
Locations (2):
- Canada (2):
  - Toronto Rehabilitation Institute, Toronto, Ontario
  - Toronto General Hospital, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: Undecided